CLINICAL TRIAL: NCT03418025
Title: Exercising Together: An Intervention for Couples Coping With Prostate Cancer During Radiation Treatment
Brief Title: Exercising Together During Radiation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00017367; NCI-2018-00031 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CPC-17135-L (Other: OHSU Knight Cancer Institute); IRB00017367 (Other: OHSU Insitutional Review Board)
Record Dates: First submitted 2018-01-24; First posted 2018-02-01 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Domestic Partnership; Prostate Carcinoma; Spouse
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Exercising Together program) (Experimental): Exercise Intervention. All participants complete questionnaires about their health status, physical activity habits and relationship with their spouse/partner and undergo four physical tests at baseline and at the end of the 5-8 week radiation treatment. The questionnaires are then completed one final time 8 weeks following the completion of radiation treatment.
  EXERCISING TOGETHER PROGRAM: Participants complete three exercise sessions (approximately 1 hour per session) per week over 5-8 weeks during radiation treatment. Participants also receive a DVD of a partnered strength training exercise program to continue on their own after radiation is completed.
  Interventions: Behavioral: Exercise Intervention; Other: Questionnaire Administration; Other: Survey Administration
- Group II (pre and post testing) (Active Comparator): Questionnaire Administration & Survey Administration. All participants complete questionnaires about their health status, physical activity habits and relationship with their spouse/partner and undergo four physical tests at baseline and at the end of the 5-8 week radiation treatment. The questionnaires are then completed one final time 8 weeks following the completion of radiation treatment.
  Interventions: Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo Exercise Together intervention
  Arms: Group I (Exercising Together program)
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well the Exercising Together program works in helping couples cope with radiation treatment for prostate cancer. Treatments for cancer can cause side effects for the patient, such as fatigue, add stress for the spousal caregiver, and put strain on the marital relationship. The Exercising Together program is designed to promote teamwork and emotional intimacy during exercise, which itself can help manage fatigue and stress for the patient and spouse, and may facilitate communication between partners about day-to-day energy, abilities, and motivation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility and acceptability of offering the Exercising Together program to couples during the time when men are undergoing an 8 week radiation treatment regimen.

SECONDARY OBJECTIVES:

I. Examine the efficacy of partnered strength training on objective physical function, self-report function, symptoms and intimacy in both the patient and his spouse.

OUTLINE:

All participants complete questionnaires about their health status, physical activity habits and relationship with their spouse/partner and undergo four physical tests at baseline and at the end of the 5-8 week radiation treatment. The questionnaires are then completed one final time 8 weeks following the completion of radiation treatment.

EXERCISING TOGETHER PROGRAM: Participants complete three exercise sessions (approximately 1 hour per session) per week over 5-8 weeks during radiation treatment. Participants also receive a digital video disc (DVD) of a partnered strength training exercise program to continue on their own after radiation is completed.

After completion of the supervised exercise program, participants are followed up at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS
* Histologically confirmed prostate cancer (confirmed by self-report on Health History Questionnaire)
* Scheduled to receive a course (5-8 weeks) of radiation treatment for prostate cancer at Oregon Health & Science University (OHSU) Department of Radiation Medicine (confirmed by self-report on Health History Questionnaire)
* Currently residing with an identifiable spouse (or co-residing partner) willing to participate (confirmed by self-report on Health History Questionnaire)
* SPOUSES
* Currently residing with the prostate cancer patient (confirmed by self-report on Health History Questionnaire)

Exclusion Criteria:

* Cognitive difficulties that preclude answering the survey questions or giving informed consent
* Medical condition, movement or neurological disorder, or medication that contraindicates participation in resistance exercise (for patient: confirmed by email and/or Electronic Privacy Information Center [EPIC] by Dr. Hung; for spouse: must answer 'No' to exercise pre-participation screening questions (question #20 & #21) in Health History Questionnaire (HHQ); if spouse answers 'Yes' to either question they will be considered eligible upon physician clearance; the exercise pre-participation screening questions are based on the American College of Sports Medicine 2016 Exercise pre-participation screening criteria)
* Currently participating in partnered strength training 2 or more times per week (confirmed by self-report on the Godin Leisure Time Exercise Questionnaire)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Feasibility | Up to 8 weeks post radiation treatment
  Will be determined as the number of couples who enroll out of those approached and the number of couples who opt to participate in Exercising Together versus to participate as controls. Will evaluate using descriptive statistics.
Physical function | Up to 8 weeks post-radiation treatment
  Will be measured by the Physical Performance Battery (PPB), developed for the Established Populations for Epidemiologic Studies of the Elderly study. The PPB consists of three timed tests: 5 repeated chair stands, standing balance, and gait speed over 4 meters. Each test is scored 0 (unable) to 4, based on quartiles of performance, then scores are summed. Higher scores indicate better physical function.
400m walk Test | Up to 8 weeks post-radiation treatment
  The 400m walk test is a self-paced, submaximal exercise test. Participants will be required to move as fast as they can along a 20m course, demarked by two cones, until they have completed 10 laps of the course (400m). The time taken to complete the test will be recorded.
Acceptability | Up to 8 weeks post-radiation treatment
  Will be measured by the average attendance at classes over the course of his radiation therapy. This will be calculated as the total number of classes attended divided by the total possible they could attend over the course of radiation therapy. Attendance will be categorized by sessions couples attended together and those where only one partner attends. Will evaluate using descriptive statistics.
Depressive symptoms | Up to 8 weeks post-radiation treatment
  Will be measured with the Center for Epidemiological Studies-Depression (CES-D) scale. Scores range from 0-60, with higher scores indicating > depressive symptomology.
Anxiety | Up to 8 weeks post-radiation treatment
  Will be measured from the Symptom Checklist - 90 Anxiety Scale (SCL-90 ANX) which includes 10 items representing anxiety symptoms, scored on a 5 point scale ranging from 0 (not at all) to 4 (extremely).
Physical intimacy | Up to 8 weeks post-radiation treatment
  Physical intimacy behavior of patient and spouse will be measured using the Physical intimacy behavior scale. Respondents are asked to report the frequency with which they engage in, initiate and avoid each of four affectionate and two sexual behaviors. Three scales assess the frequency, initiation and avoidance of affectionate and sexual behaviors.
Strain | Up to 8 weeks post-radiation treatment
  Spouse strain will be measured with the role overload scale, which assesses the extent a spouse's time and energy are exhausted by demands of care for their partner.
Dyadic coping | Up to 8 weeks post-radiation treatment
  Two types of dyadic coping will be measured. Active engagement assesses the extent to which the survivor (SVR) and spouse view their partner's active involvement and joint problem-solving. Participants respond to five items using a Likert scale from 1 (never) to 5 (very often). Higher scores indicate higher levels of perceived active engagement. Protective buffering assesses the extent to which the SVR and spouse view their partner's use of hiding concerns and denying worries. Participants respond to six items using a Likert scale from 1 (never) to 5 (very often). Higher scores indicate higher levels of perceived protective buffering.
Exercise outside the exercise intervention | Up to 8 weeks post-radiation treatment
  Will measure outside activity with the Modified Godin Leisure-Time Exercise Questionnaire (GLTEQ). This survey, reported in average minutes per week over the past month, will be broken down into four categories: mild effort (minimal effort), moderate exercise (not exhausting), and strenuous exercise (heart beats rapidly), as well as resistance (weight bearing exercise). The questionnaire will be scored three different ways, to better capture different aspects of PA: 1) total activity = vigorous + moderate + mild + resistance 2) physical activity guidelines = moderate + (vigorous x 2) 3) moderate + vigorous.
Subjective evaluation of Exercising Together Program | Up to 8 weeks post-radiation treatment
  For couples who opt to participate in Exercising Together will also ask them to fill out a survey asking about their experience in the program. They will be asked to rate their overall experience in the exercise classes using a 1 to 10 likert scale with 1 being poor and 10 being exceptional as well as indicate how much they agree or disagree with perceptions of the class.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Winters-Stone KM, Lyons KS, Beer TM, Skiba MB, Hung A. A pilot feasibility study of Exercising Together(c) during radiation therapy for prostate cancer: a dyadic approach for patients and spouses. Pilot Feasibility Stud. 2021 Dec 8;7(1):216. doi: 10.1186/s40814-021-00952-7. PMID 34879873